CLINICAL TRIAL: NCT00332306
Title: Evaluation of Safety and Efficacy of Two Different Once Daily Anti Retroviral Treatment Regimens Along With Anti-tuberculosis Treatment in Patients With HIV-1 and Tuberculosis
Brief Title: Safety and Efficacy of Two Once Daily Anti Retroviral Treatment Regimens Along With Anti-tuberculosis Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: National AIDS Control Organisation (Other); Indian Council of Medical Research (Other Government)
Responsible Party: Dr Soumya Swaminathan, Tuberculosis Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: trc23
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-01

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus Infections
Keywords: Once daily antiretroviral treatment; Concomitant antituberculosis treatment; HIV Infections
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — Didanosine; Lamivudine; efavirenz; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Didanosine + Lamivudine + Nevirapine
  Interventions: Drug: Didanosine, Lamivudine, Nevirapine
- 1 (Active Comparator): Didanosine + Lamivudine + Efavirenz
  Interventions: Drug: Didanosine, Lamivudine, Efavirenz

INTERVENTIONS:
Drug: Didanosine, Lamivudine, Efavirenz — Didanosine 250mg patients <60kg, 400mg patients > 60kg once daily Lamivudine 300 mg once daily Efavirenz 600 mg once daily All drugs will be given for 24 months
  Arms: 1
Drug: Didanosine, Lamivudine, Nevirapine — Didanosine 250 mg once daily for patients < 60kg, 400 mg OD patients > 60kg Lamivudine 300 mg once daily Nevirapine 400 mg once daily All drugs will be given for 24 months
  Arms: 2

SUMMARY:
Protocol Summary

Title: Evaluation of safety and efficacy of two different once daily anti-retroviral treatment regimens along with anti-tuberculosis treatment in patients with HIV-1 and tuberculosis - Randomized Controlled Clinical Trial

Phase: Phase III trial

Population: 180 HIV-1 positive patients with tuberculosis

Number of Sites: Four.

1. Tuberculosis Research Centre, Chennai
2. Government Medical College, Vellore
3. Government Hospital of Thoracic Medicine, Tambaram
4. Government Rajaji Hospital, Madurai

Study Duration: 26 months including 24 months of ART.

Study Objectives:

Primary Objective To compare the efficacy and safety of two different once-daily anti-retroviral treatment regimens (along with standard anti-tuberculosis treatment) in patients with HIV-1 and tuberculosis, by using virologic end points.

Secondary Objective To compare the efficacy of antiretroviral treatment given under partial supervision with unsupervised treatment (once a month supply).

DETAILED DESCRIPTION:
Description of Agent or Intervention:

The study intervention is to start patients with HIV and tuberculosis on anti-retroviral treatment along with the continuation phase of anti-tuberculosis treatment (ATT)ie after completion of first two months of treatment. The anti-TB regimen used in this trial will be 2EHRZ3/4RH3. Two different once-daily regimens are being compared for their efficacy and adverse event profile, namely ddI + 3TC + NVP versus ddI + 3TC + EFZ. The primary aim is to study the outcome of patients treated with both ART and ATT at 6 months (24 weeks of ART). A secondary objective is to compare the utility of partially supervised directly observed treatment with unsupervised administration of anti-retroviral drugs.

Patients with HIV-1 infection and active tuberculosis (pulmonary and extrapulmonary) will be started on a four-drug intermittent short-course anti-TB regimen on recruitment to the trial. They will be randomized at the end of intensive phase of ATT to receive either of the ART regimens and the outcome measured at the end of 6 months. During this phase, both ATT and ART will be given under supervision three times a week. Patients with viral load < 400 copies/ml(favourable outcome) at this time point will be randomized to receive ART either by partial observation of treatment (three times a week)or monthly supply (unsupervised administration) and final outcome will be measured at the end of 24 months of ART. The study will provide information on the comparative efficacy of the two regimens when given with anti-TB treatment as well as any added advantage that direct observation of treatment may provide.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. a) Newly diagnosed sputum smear positive tuberculosis (at least 1 out of 6 sputum specimen should be positive by smear) b)Miliary tuberculosis, mediastinal/hilar lymphadenopathy, diagnosed by chest radiography or CT scan (irrespective of sputum smear status).

   c)TB lymphadenitis with histopathological/bacteriological evidence of TB d)Pleural effusion with biochemical/cytological/bacteriological evidence of TB
3. HIV-1 positivity (on 2 different rapid tests on the same blood sample)
4. CD4 cell counts less than 250 cells/mm3
5. Likely to remain in the same area for at least two years after start of treatment.
6. Willingness to stay in the hospital for 2 weeks during initiation of ART, and attend the clinic thrice weekly for the entire period of the study (up to 2 years).
7. Willingness for home visits, and to attend for investigations, supervised treatment and follow-up as required.
8. Within the area of intake (25 kms from any of the TRC subcentres).
9. Willingness to use contraception during trial period.

Exclusion Criteria:

1. Resides outside area of intake.
2. Pregnancy and lactation.
3. Patients with major psychiatric illnesses and severe depression
4. Major complications of HIV disease like encephalopathy, renal (Serum creatinine level > 1.2 mgs/dl) or hepatic disease (Serum bilirubin > 2.0 times upper limit of normal, Serum transaminases > 2.5 times upper limit of normal), serum amylase > 2 times upper limit of normal with serum lipase > 1.5 times upper limit of normal.
5. Serious cardiac disease (CCF, IHD), uncontrolled diabetes mellitus, cancer, moribund state
6. Previous antituberculosis treatment for more than 1 month.
7. Previous antiretroviral treatment for more than 1 month
8. Patients with CD4 cell count >250 cells/mm3.
9. HIV-2 infection alone or in combination with HIV-1.
10. Patients currently using alcohol, IV drugs & other substance abuse.
11. Unwilling to use contraception & avoid pregnancy.
12. Unwilling to HIV/TB screening and participation in trial.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Suppression of Viral load to < 400 copies/ml or a two log reduction in viral load from the baseline value at the end of 6 months and a viral load <400 copies/ml at 24 months of antiretroviral therapy | Dec 2008

SECONDARY OUTCOMES:
To compare the response to treatment between partially supervised drug administration and unsupervised drug administration. | Dec 2009
To compare the tolerability and toxicity attributable to study drugs. | Dec 2009

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Swaminathan, MD, Principal Investigator — Tuberculosis Research Centre, India; PR Narayanan, PhD, Study Director — Tuberculosis Research Centre, India
Locations (1):
- Tuberculosis Research Centre, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Jack C, Lalloo U, Karim QA, Karim SA, El-Sadr W, Cassol S, Friedland G. A pilot study of once-daily antiretroviral therapy integrated with tuberculosis directly observed therapy in a resource-limited setting. J Acquir Immune Defic Syndr. 2004 Aug 1;36(4):929-34. doi: 10.1097/00126334-200408010-00006. PMID 15220699
- [Background] Patel A, Patel K, Patel J, Shah N, Patel B, Rani S. Safety and antiretroviral effectiveness of concomitant use of rifampicin and efavirenz for antiretroviral-naive patients in India who are coinfected with tuberculosis and HIV-1. J Acquir Immune Defic Syndr. 2004 Sep 1;37(1):1166-9. doi: 10.1097/01.qai.0000135956.96166.f0. PMID 15319677
- [Background] Maggiolo F, Migliorino M, Maserati R, Pan A, Rizzi M, Provettoni G, Rizzi L, Suter F; Once Study Group. Virological and immunological responses to a once-a-day antiretroviral regimen with didanosine, lamivudine and efavirenz. Antivir Ther. 2001 Dec;6(4):249-53. PMID 11878406
- [Background] Landman R, Schiemann R, Thiam S, Vray M, Canestri A, Mboup S, Kane CT, Delaporte E, Sow PS, Faye MA, Gueye M, Peytavin G, Dalban C, Girard PM, Ndoye I; Imea 011/ANRS 12-04 Study Group. Once-a-day highly active antiretroviral therapy in treatment-naive HIV-1-infected adults in Senegal. AIDS. 2003 May 2;17(7):1017-22. doi: 10.1097/00002030-200305020-00010. PMID 12700451
- [Background] Burman WJ, Jones BE. Treatment of HIV-related tuberculosis in the era of effective antiretroviral therapy. Am J Respir Crit Care Med. 2001 Jul 1;164(1):7-12. doi: 10.1164/ajrccm.164.1.2101133. No abstract available. PMID 11435232
- [Background] J. M. Molina, S Perusat, F Ferchal, C Rancinan, F raffi, W Rozenbaum, D Sereni, P Morlat, G Chene and the Montana Study Group: Once-Daily Combination Therapy with Emtricitabine, Didanosine and Efavirenz in Treatment-Naïve HIV-Infected Adults: 64-week Follow-Up of the ANRS 091 Trial.
- [Background] Ribera E, Pou L, Lopez RM, Crespo M, Falco V, Ocana I, Ruiz I, Pahissa A. Pharmacokinetic interaction between nevirapine and rifampicin in HIV-infected patients with tuberculosis. J Acquir Immune Defic Syndr. 2001 Dec 15;28(5):450-3. doi: 10.1097/00042560-200112150-00007. PMID 11744833
- [Derived] Narendran G, Menon PA, Venkatesan P, Vijay K, Padmapriyadarsini C, Ramesh Kumar S, Bhavani KP, Sekar L, Gomathi SN, Chandrasekhar C, Kumar S, Sridhar R, Swaminathan S. Acquired rifampicin resistance in thrice-weekly antituberculosis therapy: impact of HIV and antiretroviral therapy. Clin Infect Dis. 2014 Dec 15;59(12):1798-804. doi: 10.1093/cid/ciu674. Epub 2014 Aug 25. PMID 25156114
- [Derived] Swaminathan S, Padmapriyadarsini C, Venkatesan P, Narendran G, Ramesh Kumar S, Iliayas S, Menon PA, Selvaraju S, Pooranagangadevi NP, Bhavani PK, Ponnuraja C, Dilip M, Ramachandran R. Efficacy and safety of once-daily nevirapine- or efavirenz-based antiretroviral therapy in HIV-associated tuberculosis: a randomized clinical trial. Clin Infect Dis. 2011 Oct;53(7):716-24. doi: 10.1093/cid/cir447. PMID 21890776